CLINICAL TRIAL: NCT04971850
Title: Sleep-Disordered Breathing and Neurocognitive Assessment in Children and Young Adults
Acronym: TRSPed
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP210042; 2020-A03083-36 (Other: ID-RCB Number)
Record Dates: First submitted 2021-04-29; First posted 2021-07-22 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Sleep-disordered Breathing (SDB)
Keywords: Sleep-disordered breathing (SDB); Poly(somno)graphy (P(S)G); Cerebral oxygenation; Cyclic alternating pattern (CAP); Psychological and neuropsychological tests; Screening questionnaires; Treatment of SDB
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sleep-disordered breathing (SDB) (Experimental): Patients aged 1 to 20 years old with a suspicion of SDB or a high-risk of SDB due to their pathology and hospitalized at Necker Hospital for a sleep study for their clinical care.
  Interventions: Other: Sleep study

INTERVENTIONS:
Other: Sleep study — Procedures added by research during PSG :
  * SDB screening questionnaires
  * Electromyography (EMG) of accessory and abdominal muscles
  * Cerebral oxygenation
  * Mandibular movements
  * Sleep headband (pre-teens and teens) or other connected device
  * Automatic PSG analyzes
  * Psychological and neuropsychological assessment The recordings of the study will be repeated at one year if the patient needs a treatment (surgery or noninvasive ventilation) following the results of the PSG.

SUMMARY:
One of main problems in the management of sleep-disordered breathing (SDB) in children and young adults is their screening, and the absence or the weak correlation between clinical symptoms and polysomnography (PSG). It may be useful to use additional measures together with PSG to improve the detection and characterization of respiratory events during sleep and/or correlation with clinical signs of SDB.

The primary objective of the study is to determine whether psychological and neuropsychological test scores correlate with diagnostic PSG results.

DETAILED DESCRIPTION:
One of main problems in the management of sleep-disordered breathing (SDB) in children and young adults is their screening, and the absence or the weak correlation between clinical symptoms and polysomnography (PSG). It may be useful to use additional measures together with PSG to improve the detection and characterization of respiratory events during sleep and/or correlation with clinical signs of SDB.

In addition, the clinical impact of SDB and the benefit of treatment are still not clear in children and young adults, including neurocognitive and developmental perspective.

Finally, the validation of simplified tools could optimize and simplify the detection of SDB in children and young adults.

Patients scheduled to perform a diagnostic PSG for routine clinical care will have additional recordings and questionnaires as part of the study.

The primary objective of the study is to determine whether psychological and neuropsychological test scores correlate with diagnostic PSG results.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1 to 20 years with a suspicion of SDB or a high-risk of SDB due to their pathology and hospitalized at Necker Hospital for a sleep study
* Written informed consent

Exclusion Criteria:

* No social insurance
* Significant psychomotor retardation
* Cooperation not possible
* Significant agitation
* Acute condition and/or temporary drug treatments that may interfere with the results of PSG (upper or lower airway infection)
* Patient under guardianship/curatorship

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Anxiety | The day after the P(S)G
  Anxiety questionnaire using the Revised Children's Manifest Anxiety Scale (RCMAS), with an anxiety being defined by a total T-score ≥60. Mean normal value of T-score is 50 ± 10.
Depression | The day after the P(S)G
  Depression questionnaire using the Multiscore Depression Inventory for Children (MDI-C), with an abnormal score being defined by a T-score ≥70. Mean normal value of T-score is 50 ± 10.
Quality of life | The day after the P(S)G
  Quality of life questionnaire using the Pediatric Quality of Life Inventory (PedsQL). The higher the score, the better the quality of life. Min value = 0. Max value = 100.
Sensoriality | The day after the P(S)G
  Sensoriality using the Sensory profile test. Atypical performance for a raw score <122. Min value = 38. Max value = 190.
NEPSY-II memory evaluation | The day after the P(S)G
  Memory evaluation using the NEPSY-II test. Mean normal score is 10 ± 3. Abnormal for a score <4.
Children Memory Scale | The day after the P(S)G
  Memory evaluation using the Children Memory Scale test. Mean normal score is 10 ± 3. Abnormal for a score <4.
Attention | The day after the P(S)G
  Attention evaluation using the TAP test. Abnormal for a T-score <30. Mean normal value of T-score is 50 ± 10.
NEPSY-II score | The day after the P(S)G
  Executive function evaluation using the NEPSY-II. Mean normal score tests is 10 ± 3, abnormal for a score <4.
Trail Making test score | The day after the P(S)G
  Executive function evaluation using the Trail Making test. Mean normal score is 10 ± 3, abnormal for a score <4.
KiTAP subtests score | The day after the P(S)G
  Executive function evaluation using the KiTAP subtests. Abnormal T-score <30, with mean normal value of T-score is 50 ± 10.
Behavior | The day after the P(S)G
  Behavior evaluation using the Child Behaviour Checklist (CBCL). Abnormal T-score >65. Mean normal value of T-score is 50 ± 10.
Griffiths-III score | The day after the P(S)G
  Neurodevelopment evaluation using the Griffiths-III. Mean normal score is 100 ± 15. Abnormal for a score <70.
WPPSI-IV score | The day after the P(S)G
  Neurodevelopment evaluation using the WPPSI-IV. Mean normal score is 100 ± 15. Abnormal for a score <70.
WISC-V score | The day after the P(S)G
  Neurodevelopment evaluation using the WISC-V. Mean normal score is 100 ± 15. Abnormal for a score <70.
Language | The day after the P(S)G
  Language evaluation using the Griffiths-III test. Mean normal score is 100 ± 15. Abnormal for a score <70.

SECONDARY OUTCOMES:
Sleep disturbance | The day after baseline P(S)G
  Score of the sleep disturbance scale for children (SDSC) to detect the presence and severity of SDB Children < 4 years old: Min value 3, max value 15. Abnormal if score >4. Children > 4 years old: Min value 5, max value 25. Abnormal if score >12.
3D facial surface analysis | The day after baseline P(S)G
  Geometric morphometric approach based on 3D facial surface analysis of linear distances between 25 pairs of craniofacial landmarks, defined as direct Euclidean distance (in mm) between the two points.
3D facial surface analysis | The day after baseline P(S)G
  Geometric morphometric approach based on 3D facial surface analysis of geodesic distances between 25 pairs of craniofacial landmarks, defined as the shortest distance (in mm) between two points when following the contour of the face/skin.
3D facial surface analysis | The day after baseline P(S)G
  Geometric morphometric approach based on 3D facial surface analysis of angular measurements between 25 pairs of craniofacial landmarks, defined as the angles (in degree) between sets of three landmarks.
Changing detection of respiratory events | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Comparison between the apnea-hypopnea index (AHI) obtained from the P(S)G and the AHI calculated using respiratory muscle EMG
Changing detection of respiratory events | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Comparison between the AHI obtained from the P(S)G and the AHI calculated taking into account hypoventilation and flow limitation
Changing detection of respiratory events | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Comparison between the AHI obtained from the P(S)G and the AHI calculated taking into account autonomic arousals using the pulse wave amplitude
Changing detection of respiratory events | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Comparison between the AHI obtained from the P(S)G and the AHI calculated using the pulse transit time
Changing detection of respiratory events | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Comparison between the AHI obtained from the P(S)G and the AHI calculated using mandibular movements
Changing detection of respiratory events | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Comparison between the AHI obtained from the P(S)G and the AHI calculated using cerebral oxygenation desaturations
Correlations with clinical signs of SDB | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between clinical signs by questionnaire and respiratory muscles power by EMG.
Correlations with clinical signs of SDB | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between clinical signs by questionnaire and hypoventilation and flow limitation scores by P(S)G.
Correlations with clinical signs of SDB | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between clinical signs by questionnaire and autonomic arousals using pulse wave amplitude by pulse oximetry.
Correlations with clinical signs of SDB | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between clinical signs by questionnaire and pulse transit time analysis by ECG.
Correlations with clinical signs of SDB | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between clinical signs by questionnaire and mandibular movement analysis by non-invasive magnetic distance sensors.
Correlations with clinical signs of SDB | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between clinical signs by questionnaire and cerebral oxygenation analysis by near-infrared spectroscopy.
Correlations with clinical signs of SDB | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between clinical signs by questionnaire and the type of CAP by EEG.
Correlations with pulse oximetry | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between pulse oximetry and respiratory muscles power by EMG.
Correlations with pulse oximetry | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between pulse oximetry and hypoventilation and flow limitation scores by P(S)G.
Correlations with pulse oximetry | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between pulse oximetry and autonomic arousals using pulse wave amplitude.
Correlations with pulse oximetry | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between pulse oximetry and pulse transit time analysis.
Correlations with pulse oximetry | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between pulse oximetry and mandibular movement analysis by non-invasive magnetic distance sensors.
Correlations with pulse oximetry | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between pulse oximetry and cerebral oxygenation analysis by near-infrared spectroscopy.
Correlations with pulse oximetry | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between pulse oximetry and the type of CAP.
Correlations with sleep questionnaires | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between sleep questionnaires and respiratory muscles EMG.
Correlations with sleep questionnaires | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between sleep questionnaires and hypoventilation and flow limitation scores by P(S)G.
Correlations with sleep questionnaires | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between sleep questionnaires and autonomic arousals using pulse wave amplitude.
Correlations with sleep questionnaires | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between sleep questionnaires and pulse transit time analysis.
Correlations with sleep questionnaires | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between sleep questionnaires and mandibular movement analysis by non-invasive magnetic distance sensors.
Correlations with sleep questionnaires | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between sleep questionnaires and cerebral oxygenation analysis.
Correlations with sleep questionnaires | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between sleep questionnaires and the type of CAP.
Correlations with psychological and neuropsychological tests | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between psychological and neuropsychological scores and the different calculated AHI.
Correlations with psychological and neuropsychological tests | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between psychological and neuropsychological scores and the types of CAP.
Correlations with psychological and neuropsychological tests | The day after baseline P(S)G and 1 year after the intervention/procedure/surgery
  Correlation between psychological and mean nocturnal cerebral oxygenation.
Alternative analysis | The day after baseline P(S)G
  Correlation between the AHI obtained from P(S)G and the AHI obtained using respiratory inductance plethysmography.
Alternative analysis in (pre-)teens | The day after baseline P(S)G
  Correlations between sleep stages obtained from PSG and sleep stages from a sleep headband.
Alternative analysis | The day after baseline P(S)G
  Correlations between the sleep stages and AHI obtained from manual analysis of PSG and an automatic analysis.
Effect of treatment on Griffiths-III score | At one year
  Comparison of neurodevelopment evaluation using the Griffiths-III between baseline and 1 year following treatment for severe or moderate-to-severe (pubescent patient) obstructive sleep apnea. Mean normal score is 100 ± 15. Abnormal for a score <70.
Effect of treatment on WPPSI-IV score | At one year
  Comparison of neurodevelopment evaluation using the WPPSI-IV between baseline and 1 year following treatment for severe or moderate-to-severe (pubescent patient) obstructive sleep apnea. Mean normal score is 100 ± 15. Abnormal for a score <70.
Effect of treatment on WISC-V score | At one year
  Comparison of neurodevelopment evaluation using the WISC-V between baseline and 1 year following treatment for severe or moderate-to-severe (pubescent patient) obstructive sleep apnea. Mean normal score is 100 ± 15. Abnormal for a score <70.
Effect of treatment | At one year
  Comparison of the percentage of types of CAP between baseline and 1 year following treatment.
Effect of treatment | At one year
  Comparison of mean cerebral oxygenation between baseline and 1 year following treatment.
Effect of treatment on Pittsburgh Sleep Quality Index (PSQI) | At one year
  Comparison of PSQI scores between baseline and 1 year following treatment. PSQI max score = 21. Threshold values for the PSQI scale: 0-4: Good, 5-8: Moderate, >9: Bad sleep quality.
Effect of treatment on Epworth sleepiness scale (ESS) | At one year
  Comparison of ESS scores between baseline and 1 year following treatment. ESS max score = 33. Threshold values for the ESS scale: <8: No, 9-14: Moderate, >15: Severe sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Fauroux, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Sonia Khirani, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No